CLINICAL TRIAL: NCT00476320
Title: The Use of Myocardial Deformation Imaging Based on Ultrasonic Pixel Tracking to Identify Reversible Myocardial Dysfunction
Brief Title: The Use of Myocardial Deformation Imaging
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Other Study IDs: Becker-LE-FU-2007
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Myocardial Viability in Ischemic Left Ventricular Dysfunction; Prediction for Improvement in Cardiac Function After Revascularization Therapy
Keywords: echocardiography; myocardial infarction; magnetic resonance imaging; revascularization; viability
MeSH Terms: conditions — Myocardial Infarction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging
Procedure: Revascularization
Procedure: Echocardiography with myocardial deformation imaging

SUMMARY:
Myocardial deformation imaging allows analysis of myocardial viability in ischemic left ventricular dysfunction. This study will evaluate the predictive value of myocardial deformation imaging for improvement in cardiac function after revascularization therapy in comparison to contrast-enhanced cardiac magnetic resonance imaging (ceMRI).

In 55 patients with ischemic left ventricular dysfunction, myocardial viability was assessed using pixel-tracking-derived myocardial deformation imaging and ceMRI to predict recovery of function at 9±2 months follow-up. For each left ventricular segment in a 16-segment model peak systolic radial strain will be determined from parasternal 2D echocardiographic views and the amount of late hyperenhancement (LE) and maximal thickness of myocardial tissue without LE using ceMRI. The hypothesis is that compared with segments showing functional improvement, those that failed to recover had lower radial strain and lower thickness without LE and higher LE.

DETAILED DESCRIPTION:
Between August 2004 and June 2006 195 patients with ischemic left ventricular dysfunction underwent MRI for the definition of myocardial viability. Onehundred-ten patients with non-ischemic cardiomyopathy or acute coronary syndromes were excluded from the study to avoid possible acute ischemia or stunning. Within the 85 patients with chronic ischemic heart disease, six patients refused participation in this study and five patients had echocardiographic windows insufficient for participation. Within the remaining 74 patients 55 patients underwent revascularization and 19 had no revascularization. These 55 patients form our study group! Functional recovery will be assessed using echocardiographic images before and 9±2 months after revascularization with a Vivid Seven System (GE Vingmed, Horton, Norway). Parasternal long-axis and short-axis views at basal, midventricular and apical levels, as well as 3 standard apical views (4 chamber, 2 chamber, and long axis) have been acquired (frame rate 56 to 92 frames/s). Segmental wall motion will be determined using the following score: 1=normokinetic, 1.5= mildly hypokinetic, 2= moderately or severely hypokinetic, 3= akinetic, or 4= dyskinetic. A segment is considered to demonstrate functional improvement during follow-up if it improved by at least 1 grade. Global functional recovery was considered in case of an increase in ejection fraction>5% at follow-up.

The three acquired parasternal short axis views will be analysed with the aid of a dedicated software package (EchoPAC BT 05.2, GE Vingmed, Horton, Norway). This system allows analysis of peak systolic circumferential and radial strain from short axis views based on detection of natural acoustic markers. The system calculates mean strain values for whole predefined LV segments, including all myocardial layers from the endocardium to epicardium.

All patients underwent cMRI within a few hours of the baseline echocardiographic study on a 1.5-T whole-body MR scanner (Intera, Best, Philips, the Netherlands). The assignment to a hyperenhancement category reflects the extent of hyperenhancement within each segment by visual assessment considering a 5-group scale: 0% hyperenhancement (group 1), 1 to 25% hyperenhancement (group 2), 26 to 50% hyperenhancement (group 3), 51 to 75% hyperenhancement (group 4) and 76 to 100% hyperenhancement (group 5).

In addition, the maximal thickness of myocardial tissue without late hyperenhancement will be determined for each LV segment. This is considered to be a parameter of the remaining viable myocardium.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic left ventricular dysfunction scheduled for coronary revascularization

Exclusion Criteria:

* Patients with acute coronary syndrome and poor echocardiographic windows

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-08; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Becker, PhD, MD, Principal Investigator — RWTH Aachen University Hospital; Rainer Hoffmann, Professor, Study Chair — RWTH Aachen University Hospital; Malte Kelm, Professor, Study Director — RWTH Aachen University Hospital
Locations (1):
- RWTH University Hospital, Aachen, Germany

REFERENCES:
- [Result] Becker M, Hoffmann R, Kuhl HP, Grawe H, Katoh M, Kramann R, Bucker A, Hanrath P, Heussen N. Analysis of myocardial deformation based on ultrasonic pixel tracking to determine transmurality in chronic myocardial infarction. Eur Heart J. 2006 Nov;27(21):2560-6. doi: 10.1093/eurheartj/ehl288. Epub 2006 Oct 11. PMID 17035253
- [Result] Kim RJ, Wu E, Rafael A, Chen EL, Parker MA, Simonetti O, Klocke FJ, Bonow RO, Judd RM. The use of contrast-enhanced magnetic resonance imaging to identify reversible myocardial dysfunction. N Engl J Med. 2000 Nov 16;343(20):1445-53. doi: 10.1056/NEJM200011163432003. PMID 11078769
- [Result] Reisner SA, Lysyansky P, Agmon Y, Mutlak D, Lessick J, Friedman Z. Global longitudinal strain: a novel index of left ventricular systolic function. J Am Soc Echocardiogr. 2004 Jun;17(6):630-3. doi: 10.1016/j.echo.2004.02.011. PMID 15163933
- [Derived] Becker M, Altiok E, Lente C, Otten S, Friedman Z, Adam D, Hoffmann R, Koos R, Krombach G, Marx N, Hoffmann R. Layer-specific analysis of myocardial function for accurate prediction of reversible ischaemic dysfunction in intermediate viability defined by contrast-enhanced MRI. Heart. 2011 May;97(9):748-56. doi: 10.1136/hrt.2010.210906. Epub 2011 Mar 17. PMID 21415076
- [Derived] Becker M, Lenzen A, Ocklenburg C, Stempel K, Kuhl H, Neizel M, Katoh M, Kramann R, Wildberger J, Kelm M, Hoffmann R. Myocardial deformation imaging based on ultrasonic pixel tracking to identify reversible myocardial dysfunction. J Am Coll Cardiol. 2008 Apr 15;51(15):1473-81. doi: 10.1016/j.jacc.2007.10.066. PMID 18402903